CLINICAL TRIAL: NCT00573989
Title: Phase I/II Clinical Trial of Combined Pre-Irradiation With Pemetrexed and Erlotinib Followed by Maintenance Erlotinib for Recurrent and Second Primary Squamous Cell Carcinoma of the Head and Neck
Brief Title: Intensity-Modulated Radiation Therapy, Pemetrexed, and Erlotinib in Treating Patients With Recurrent or Second Primary Head and Neck Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Drug Supply Issue
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00003457; P30CA012197 (NIH); CCCWFU-60107; NCT01580449 (obsolete NCT alias)
Record Dates: First submitted 2007-12-13; First posted 2007-12-14 (Estimated); Results first posted 2018-12-13 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2018-12

CONDITIONS: Head and Neck Cancer
Keywords: recurrent squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the larynx; recurrent verrucous carcinoma of the larynx; recurrent squamous cell carcinoma of the lip and oral cavity; recurrent verrucous carcinoma of the oral cavity; metastatic squamous neck cancer with occult primary squamous cell carcinoma; recurrent metastatic squamous neck cancer with occult primary; recurrent squamous cell carcinoma of the oropharynx
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Erlotinib Hydrochloride; Pemetrexed; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Erlotinib (Experimental): Erlotinib
  Interventions: Drug: erlotinib hydrochloride; Drug: pemetrexed disodium; Procedure: quality-of-life assessment; Radiation: intensity-modulated radiation therapy

INTERVENTIONS:
Drug: erlotinib hydrochloride
Drug: pemetrexed disodium
Procedure: quality-of-life assessment
Radiation: intensity-modulated radiation therapy

SUMMARY:
RATIONALE: Specialized radiation therapy that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue. Drugs, such as pemetrexed and erlotinib, may make tumor cells more sensitive to radiation therapy. Erlotinib and pemetrexed may also stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving intensity-modulated radiation therapy together with pemetrexed and erlotinib may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of erlotinib when given together with intensity-modulated radiation therapy and pemetrexed and to see how well they work in treating patients with recurrent or second primary head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the acute toxicity and feasibility of intensity modulated radiotherapy (IMRT) in combination with radiosensitizing drugs pemetrexed disodium and erlotinib hydrochloride in patients with recurrent or second primary squamous cell carcinoma of the head and neck. (Phase I)
* Determine the maximum tolerated dose and recommended phase II dose of erlotinib hydrochloride in these patients. (Phase I)
* Determine progression-free survival (PFS) at 1 year in these patients. (Phase II)

Secondary

* Determine median PFS, median overall survival (OS), and OS at 1 and 2 years in these patients.
* Determine objective tumor response as measured by CT scan or MRI in these patients.
* Evaluate the acute and chronic toxicity of IMRT in combination with radiosensitizing drugs pemetrexed disodium and erlotinib hydrochloride in these patients.
* Evaluate the impact of treatment on quality of life as measured by FACT-H&N, PSS-HN, MD Anderson Dysphagia Inventory (MDADI), and swallowing by direct functional measurements at different time points.
* Evaluate the level of phosphorylation of different tyrosine residues within the cytoplasmic domain of EGFR, bound adaptors, as well as markers of downstream pathways activation by nano LC-MS/MS in tumor tissue and correlate with levels of P-AKT and P-ERK by immunohistochemistry and with response to treatment.
* Measure the levels of TS and p53 and correlate with treatment response.

OUTLINE: This is a phase I, dose-escalation study of erlotinib hydrochloride followed by a phase II study.

* Phase I: Patients undergo intensity modulated radiotherapy (IMRT) once daily, 5 days a week, for 6 weeks. Patients receive pemetrexed disodium IV over 10 minutes on day 1 of radiotherapy. Treatment with pemetrexed disodium repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity. Patients also receive oral erlotinib hydrochloride once daily beginning on day 1 of radiotherapy and continuing for up to 2 years in the absence of disease progression or unacceptable toxicity.
* Phase II: Patients undergo IMRT and receive pemetrexed sodium as in phase I. Patients also receive erlotinib hydrochloride at the maximum tolerated dose determined in phase I.

Quality of life is assessed at baseline, weekly during treatment, at 1, 6, and 12 months, and then annually thereafter.

After completion of study treatment, patients are followed every 3 months for 2 years, every 6 months for 1 year, and then annually thereafter.

ELIGIBILITY:
Inclusion:

* Histologically or cytologically confirmed diagnosis of recurrent or second primary squamous cell carcinoma (SCC) of the head and neck, including any of the following:

* Oral cavity
* Oropharynx
* Hypopharynx
* Larynx
* Recurrent neck metastases with unknown primary

Exception from pathology confirmation of tumor recurrence is accepted for patients who originally had pathologically confirmed SCC of the Head and Neck, the new tumor is located in the head and neck area and it is clinically considered as a recurrence of the original tumor, and a tumor biopsy is technically difficult and would expose the patient to unjustified risk. The treating physicians should agree and document the clinical definition of tumor recurrence and should document the increased risk for biopsy.

* Measurable disease by CT scan or MRI OR evaluable disease
* No definitive evidence of distant metastasis
* Unresectable disease by a preliminary ENT evaluation OR refused surgery
* Patients may have received chemotherapy as a component of their primary tumor treatment but not for recurrent or metastatic disease. No prior treatment with systemic anti-EGFR inhibitors or Pemetrexed is permitted
* Has undergone prior head and neck radiotherapy (for SCC of the head and neck) to a dose of ≤ 72 Gy that involved most of the recurrent tumor (> 75%) OR has a second primary tumor volume in areas previously irradiated to > 45 Gy
* The entire tumor volume must be included in a treatment field that limits the total spinal cord dose to 54 Gy (prior plus planned dose)
* Must have disease recurrence or persistence for ≥ 6 months after completion of prior radiotherapy
* ECOG performance status 0-1
* Age ≥ 18 years
* ANC > 1,500/µL
* Platelet count > 100,000/µL
* Total bilirubin < 1.5 times upper limit of normal (ULN)
* AST/ALT < 2 times ULN
* Creatinine < 1.5 times ULN
* Willing and able to take folic acid and vitamin B12 supplementation
* Recovered from prior surgery, chemotherapy, or radiotherapy
* At least 6 months since prior radiotherapy
* At least 5 days since prior aspirin or other non-steroidal anti-inflammatory agents (8 days for long acting agents [e.g., piroxicam])
* Fertile patients must use effective contraception

Exclusion:

* Nasopharyngeal carcinoma
* Concurrent uncontrolled illness, including, but not limited to, any of the following:

  * Ongoing or active infection
  * Psychiatric illness or social situation that would limit compliance with study requirements
  * Significant history of uncontrolled cardiac disease (i.e., uncontrolled hypertension; unstable angina; recent myocardial infarction [within the past 3 months]; uncontrolled congestive heart failure; or cardiomyopathy with decreased ejection fraction)
* Active interstitial lung disease
* Presence of third space fluid that cannot be controlled by drainage
* Other concurrent investigational agents
* Pregnant or nursing
* HIV positive

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2008-03 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mercedes Porosnicu, MD, Principal Investigator — Wake Forest University Health Sciences; Kathryn M. Greven, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (2):
- United States (2):
  - UNC Linberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina

RESULTS

PARTICIPANT FLOW:
Groups:
- Erlotinib 100mg: Participants will be given 100mg of erlotinib, pemetrexed disodium, and intensity-modulated radiation therapy.
- Erlotinib 125mg: Participants will be given 125mg of erlotinib, pemetrexed disodium, and intensity-modulated radiation therapy.
- Erlotinib 150mg: Participants will be given 150mg of erlotinib, pemetrexed disodium, and intensity-modulated radiation therapy.
- Erlotinib 125mg- Phase II: Participants in phase II will be given 125mg of erlotinib, pemetrexed disodium, and intensity-modulated radiation therapy.
Period: Erlotinib Phase I
Arm/Group | Erlotinib 100mg | Erlotinib 125mg | Erlotinib 150mg | Erlotinib 125mg- Phase II
Started | 4 | 6 | 5 | 0
Completed | 4 | 6 | 5 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Erlotinib 125mg- Phase II
Arm/Group | Erlotinib 100mg | Erlotinib 125mg | Erlotinib 150mg | Erlotinib 125mg- Phase II
Started | 0 | 0 | 0 | 12
Completed | 0 | 0 | 0 | 12
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Combined Re-irradiation With Pemetrexed And Erlotinib Followed by Maintenance Erlotinib
Groups:
- Erlotinib: Erlotinib
  erlotinib hydrochloride
  pemetrexed disodium
  quality-of-life assessment
  intensity-modulated radiation therapy
Arm/Group | Erlotinib
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.96 (7.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 25
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of Erlotinib Hydrochloride (Phase I)
Description: Dose at which 100% of participants tolerated the dose
Time Frame: 56 Days
Measure: Number; unit: mg
Arm/Group | Erlotinib
Number analyzed (Participants) | 27
mg | 125

2. Primary Outcome: Progression-free Survival (PFS) at 1 Year (Phase II)
Description: Determine Progression Free Survival at 1 year defined as the percentage of patients who are alive at 1 year after beginning of their concurrent re-irradiation and chemotherapy without loco-regional progression of their disease as measured by CT scan or MRI.
Time Frame: 1 year
Population: Data corresponds to Phase II patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Erlotinib
Number analyzed (Participants) | 12
Participants | 5

3. Secondary Outcome: Median Progression Free Survival
Description: Median Progression Free Survival of participants reported after 2 years.
Time Frame: 2 years
Population: Data corresponds to Phase II patients.
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Erlotinib
Number analyzed (Participants) | 12
years | .71 [.58 to .99]

4. Secondary Outcome: Median Overall Survival
Description: Median Overall Survival of participants reported after 2 years.
Time Frame: up to 5 years
Population: Data corresponds to Phase II patients.
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Erlotinib
Number analyzed (Participants) | 12
years | 1.01 [.65 to 3.08]

5. Secondary Outcome: Overall Survival
Description: Overall survival of participants reported after 2 years.
Time Frame: 1 and 2 years
Population: Data corresponds to Phase II patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Erlotinib
Number analyzed (Participants) | 12
Participants
  1 year | 9
  2 years | 7

6. Secondary Outcome: Evaluation of Acute and Chronic Toxicity
Description: Evaluate acute and chronic toxicity of the combined re-irradiation with radiosensitizing drugs: Pemetrexed and Erlotinib. Adverse events with Common Toxicity Criteria grades of 4 and 5 are reported for phase I and II.
Time Frame: 1 year
Measure: Number; unit: events
Arm/Group | Erlotinib
Number analyzed (Participants) | 25
events
  phase I | 18
  phase II | 6

7. Secondary Outcome: Change in Quality of Life- FACT H&N
Description: The Functional Assessment of Cancer Therapy-Head and Neck (FACT H&N) consists of 27 core items which assess patient function in four domains: Physical, Social/Family, Emotional, and Functional well-being, which is further supplemented by 12 site specific items to assess for head and neck related symptoms. Each item is rated on a 0 to 4 Likert type scale, and then combined to produce subscale scores for each domain. Score range is 0-156. Higher scores denotes better outcomes
Time Frame: baseline and 12 months
Population: Data not collected for all participants at 12 months. Data corresponds to Phase II patients.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Erlotinib
Number analyzed (Participants) | 10
units on a scale
  baseline | 84.87 (8.19)
  12 months: number analyzed (Participants) | 3
  12 months | 88.61 (18.64)

8. Secondary Outcome: Change in Quality of Life: PSS-HN
Description: The Performance Status Scale for Head & Neck Cancer Patients (PSS-HN) is s designed to evaluate performance in areas of functioning most likely affected by head and neck cancer and its treatment, specifically Normalcy of Diet, Eating in Public, and Understandability of Speech. Each subscale is rated from 0 to 100, with higher scores indicating better performance
Time Frame: baseline and 6 months
Population: Data not collected for all participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Erlotinib
Number analyzed (Participants) | 9
units on a scale
  Eating Baseline: number analyzed (Participants) | 8
  Eating Baseline | 56.25 (34.72)
  Eating 6 months: number analyzed (Participants) | 4
  Eating 6 months | 43.75 (23.94)
  Speech Baseline: number analyzed (Participants) | 8
  Speech Baseline | 81.25 (11.57)
  Speech 6 months: number analyzed (Participants) | 4
  Speech 6 months | 75.0 (20.41)
  Diet Baseline | 44.44 (44.47)
  Diet 6 months: number analyzed (Participants) | 4
  Diet 6 months | 25.0 (50.0)

9. Secondary Outcome: Change in Quality of Life: MDADI
Description: The M.D. Anderson Dysphagia Inventory (MDADI) was used to assess effects of dysphagia on the quality of life of patients with head and neck cancer. It incorporates 3 domains (emotional, functional, and physical) as well as 1 global question. Each subscale with five possible responses scored on a scale of 1 to 5 (strongly agree, agree, no opinion, disagree and strongly disagree). Scores range from 0 (extremely low functioning) to 100 (higher functioning). Higher MDADI score represents better day-to-day functioning and better quality of life.
Time Frame: baseline and 12 months
Population: Data not collected on all participants at 12 months. Data corresponds to Phase II patients.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Erlotinib
Number analyzed (Participants) | 9
units on a scale
  baseline- global | 64.44 (26.03)
  12 months- global: number analyzed (Participants) | 2
  12 months- global | 90.0 (14.14)
  baseline- emotion | 70.37 (9.2)
  12 months- emotion: number analyzed (Participants) | 2
  12 months- emotion | 78.33 (2.36)
  baseline- function | 65.78 (12.98)
  12 months- function: number analyzed (Participants) | 2
  12 months- function | 84.0 (5.66)
  baseline- physical | 60.0 (7.91)
  12 months- physical: number analyzed (Participants) | 2
  12 months- physical | 73.75 (8.84)

10. Secondary Outcome: Evaluation of Biomarkers
Time Frame: throughout study completion, up to 2 years
Population: Patients refused biopsy, so no data collected.
Arm/Group | Erlotinib
Number analyzed (Participants) | 0

11. Secondary Outcome: Objective Tumor Response
Description: Objective Tumor Response reported on participants at 1 year (complete, partial, progression, or stable response).
Time Frame: 1 year
Population: Data corresponds to Phase II patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Erlotinib
Number analyzed (Participants) | 12
Participants
  Complete | 7
  Partial | 5
  Progression | 4
  Stable | 2

ADVERSE EVENTS:
Time Frame: up to 5 years
Description: All-Cause Mortality data was collected for all 12 participants in the "Erlotinib 125mg Phase II" Arm/Group, while Serious Adverse Events and Other (Not Including Serious) Adverse Events data were only collected for 11 participants in this Arm/group
Groups:
- Erlotinib 100 mg: Participants will be given 100mg of erlotinib, pemetrexed disodium, and intensity-modulated radiation therapy.
- Erlotinib 125mg Phase II: Participants in phase II will be given 125mg of erlotinib, pemetrexed disodium, and intensity-modulated radiation therapy.
Arm/Group | Erlotinib 100 mg | Erlotinib 125mg | Erlotinib 150mg | Erlotinib 125mg Phase II
All-Cause Mortality (participants affected / at risk) | 4/4 | 6/6 | 5/5 | 8/12
Serious Adverse Events (participants affected / at risk) | 3/4 | 6/6 | 5/5 | 5/11
Other Adverse Events (participants affected / at risk) | 4/4 | 6/6 | 5/5 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib 100 mg (N=4) | Erlotinib 125mg (N=6) | Erlotinib 150mg (N=5) | Erlotinib 125mg Phase II (N=11)
Hypoxia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Neutrophils/granulocytes (Immune system disorders) | 1 | 1 | 1 | 1 — (ANC/AGC) 1.6-7.3
Obstruction/stenosis of airway (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 — Trachea
CPK (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 — creatine phosphokinase
Calcium, serum-low (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 — hypocalcemia
Cardiac ischemia/infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac troponin I (Cardiac disorders) | 0 | 1 | 0 | 0 — cTnI
Cardiopulmonary arrest, cause unknown (Cardiac disorders) | 0 | 1 | 0 | 0 — non-fatal
Leukocytes (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1 — (total WBC) (4.8-10.8)
Pain (Cardiac disorders) | 0 | 1 | 0 | 0 — Cardiac/heart
Acidosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 — (metabolic or respiratory) (7.35-7.45)
Gastrointestinal (Gastrointestinal disorders) | 0 | 0 | 1 | 0 — Other
Hemoglobin (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 — (gender based)
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 — (1-5.1)
Hemorrhage, pulmonary/upper respiratory (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 — Bronchopulmonary NOS
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib 100 mg (N=4) | Erlotinib 125mg (N=6) | Erlotinib 150mg (N=5) | Erlotinib 125mg Phase II (N=11)
ALT, SGPT (Hepatobiliary disorders) | 3 | 4 | 3 | 3 — (serum glutamic pyruvic transaminase) ((2 -50)
AST, SGOT (Hepatobiliary disorders) | 1 | 4 | 4 | 4 — (serum glutamic oxaloacetic transaminase) (5-40)
Albumin, serum-low (Blood and lymphatic system disorders) | 3 | 6 | 5 | 8 — (hypoalbuminemia) (3.5-5.0)
Alkaline phosphatase (General disorders) | 1 | 3 | 1 | 3 — (25-125)
Allergic rhinitis (Immune system disorders) | 2 | 0 | 0 | 1 — (including sneezing, nasal stuffiness, postnasal drip)
Anorexia (Metabolism and nutrition disorders) | 0 | 4 | 2 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 — (non-septic)
Bilirubin (Blood and lymphatic system disorders) | 3 | 4 | 3 | 5 — (hyperbilirubinemia) (0.1-1.2)
Calcium, serum-low (Blood and lymphatic system disorders) | 3 | 4 | 5 | 9 — (hypocalcemia)
Cardiac General (Cardiac disorders) | 0 | 0 | 0 | 1 — Other
Cervical spine (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 — range of motion
Constipation (Gastrointestinal disorders) | 2 | 2 | 2 | 5
Cough (General disorders) | 2 | 3 | 1 | 4
Creatinine (Blood and lymphatic system disorders) | 0 | 2 | 2 | 2 — (0.5-1.5)
Dehydration (General disorders) | 1 | 2 | 3 | 6
Dermatology/Skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 4 | 2 | 8
Dizziness (General disorders) | 2 | 0 | 1 | 2
Dry eye syndrome (Eye disorders) | 2 | 0 | 0 | 1
Dry mouth/salivary gland (General disorders) | 0 | 2 | 0 | 1 — (xerostomia)
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 2
Dysphagia (General disorders) | 3 | 1 | 2 | 7 — (difficulty swallowing)
Edema (General disorders) | 1 | 1 | 1 | 1 — head and neck
Esophagitis (General disorders) | 1 | 0 | 0 | 1
Eyelid dysfunction (Eye disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 3 | 4 | 8 — (asthenia, lethargy, malaise)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 — (fever of unknown origin without clinically or microbiologically documented infection)(ANC <1.0 x 10e9/L, fever >=38.5 degrees C)
Fever (General disorders) | 1 | 3 | 2 | 1 — (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L)
Fistula, GI (Gastrointestinal disorders) | 0 | 0 | 0 | 1 — Pharynx
Gastritis (Gastrointestinal disorders) | 1 | 1 | 0 | 2 — (including bile reflux gastritis)
Gastrointestinal - Other (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Glucose, serum-high (Blood and lymphatic system disorders) | 3 | 5 | 4 | 10 — (hyperglycemia)
Glucose, serum-low (Blood and lymphatic system disorders) | 2 | 0 | 1 | 3 — (hypoglycemia)
Hearing (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 — patients without baseline audiogram and not enrolled in a monitoring program
Hemoglobin (Blood and lymphatic system disorders) | 4 | 6 | 4 | 10 — (gender based)
Hemorrhage, pulmonary/upper respiratory (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Hypertension (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Hypotension (Blood and lymphatic system disorders) | 1 | 3 | 3 | 1
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 1 | 0 | 0 | 1 — Lip/perioral
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 0 | 0 | 0 | 1 — Middle ear (otitis media)
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 1 | 2 | 0 | 2 — Skin (cellulitis)
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 0 | 0 | 0 | 1 — Urinary tract NOS
Infection with unknown ANC (Infections and infestations) | 0 | 0 | 0 | 1 — Foreign body (e.g., graft, implant, prosthesis, stent)
Infection with unknown ANC (Infections and infestations) | 1 | 0 | 1 | 2 — Lung (pneumonia)
Infection with unknown ANC (Infections and infestations) | 0 | 0 | 0 | 1 — Neck NOS
Infection with unknown ANC (Infections and infestations) | 0 | 0 | 0 | 2 — Upper airway NOS
Insomnia (Nervous system disorders) | 0 | 0 | 0 | 1
Leukocytes (Blood and lymphatic system disorders) | 4 | 4 | 4 | 10 — (total WBC) (4.8-10.8)
Lymphedema-related fibrosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 4 | 6 | 4 | 10 — (1-5.1)
Magnesium, serum-high (Renal and urinary disorders) | 2 | 3 | 1 | 3 — (hypermagnesemia)
Magnesium, serum-low (Renal and urinary disorders) | 2 | 3 | 3 | 5 — (hypomagnesemia)
Mood alteration (Nervous system disorders) | 0 | 1 | 1 | 3 — Anxiety
Mood alteration (Nervous system disorders) | 0 | 0 | 0 | 2 — Depression
Mucositis/stomatitis (clinical exam) (General disorders) | 1 | 0 | 0 | 2 — Larynx
Mucositis/stomatitis (clinical exam) (General disorders) | 2 | 3 | 1 | 9 — Oral cavity
Musculoskeletal/Soft Tissue - Other (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 5 | 4 | 8
Neutrophils/granulocytes (Immune system disorders) | 1 | 3 | 3 | 5 — (ANC/AGC) 1.6-7.3
Pain: Abdomen NOS (Musculoskeletal and connective tissue disorders) | 2 | 0 | 3 | 2
Pain: Chest/thorax NOS (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2
Pain: Eye (Eye disorders) | 1 | 0 | 0 | 1
Pain: Head/headache (General disorders) | 2 | 0 | 0 | 2
Pain: Neck (General disorders) | 1 | 3 | 1 | 2
Pain: Oral cavity (General disorders) | 0 | 1 | 1 | 3
Pain: Oral-gums (General disorders) | 0 | 0 | 0 | 1
Pain: Scalp (General disorders) | 1 | 0 | 0 | 1
Pain: Stomach (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Pain: Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 1
Phosphate, serum-low (Blood and lymphatic system disorders) | 2 | 1 | 2 | 1 — (hypophosphatemia)
Platelets (Blood and lymphatic system disorders) | 2 | 4 | 3 | 7 — (160-360)
Potassium, serum-high (hyperkalemia) (3.5-5.3) (Blood and lymphatic system disorders) | 1 | 1 | 1 | 5
Potassium, serum-low (hypokalemia) (3.5-5.3) (Blood and lymphatic system disorders) | 2 | 3 | 4 | 3
Pulmonary/Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 3 | 3 | 4 | 4
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1 | 3 | 2 | 5
Rash: dermatitis associated with radiation: Chemoradiation (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 3
Rash: dermatitis associated with radiation: Radiation (Skin and subcutaneous tissue disorders) | 0 | 5 | 1 | 4
Rigors/chills (General disorders) | 0 | 0 | 0 | 1
Skin breakdown/decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Sodium, serum-high (Renal and urinary disorders) | 0 | 0 | 1 | 3 — (hypernatremia) (135-146)
Sodium, serum-low (Renal and urinary disorders) | 4 | 4 | 2 | 7 — (hyponatremia) (135-146)
Supraventricular and nodal arrhythmia: Atrial tachycardia/Paroxysmal Atrial Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 1
Supraventricular and nodal arrhythmia: Sinus bradycardia (Cardiac disorders) | 2 | 1 | 0 | 1
Supraventricular and nodal arrhythmia: Sinus tachycardia (Cardiac disorders) | 2 | 1 | 0 | 1
Sweating (diaphoresis) (General disorders) | 0 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Trismus (difficulty, restriction or pain when opening mouth) (General disorders) | 2 | 0 | 0 | 1
Vision-flashing lights/floaters (Eye disorders) | 0 | 0 | 0 | 1
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2 | 3 | 4
Weight loss (General disorders) | 1 | 1 | 0 | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0
Bone (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 — spine-scoliosis
Distension/bloating, abdominal (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 2 | 0 — (shortness of breath)
Edema: limb (General disorders) | 1 | 2 | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Heartburn/dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Hemorrhage, pulmonary/upper respiratory: Pharynx (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hemorrhage, pulmonary/upper respiratory: Respiratory tract NOS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hemorrhage, pulmonary/upper respiratory: Stoma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hemorrhage, pulmonary/upper respiratory: Trachea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hemorrhage/Bleeding - Other (General disorders) | 1 | 0 | 0 | 0
Hypoxia (Blood and lymphatic system disorders) | 0 | 1 | 2 | 1
Infection with normal ANC or Grade 1 or 2 neutrophils: Conjunctiva (Infections and infestations) | 1 | 1 | 0 | 0
Infection with normal ANC or Grade 1 or 2 neutrophils: Trachea (Infections and infestations) | 1 | 2 | 0 | 0
Infection with normal ANC or Grade 1 or 2 neutrophils: Vagina (Infections and infestations) | 1 | 0 | 0 | 0
Infection with unknown ANC: Conjunctiva (Infections and infestations) | 1 | 0 | 0 | 0
Infection with unknown ANC: Lip/perioral (Infections and infestations) | 1 | 0 | 0 | 0
Infection with unknown ANC: Skin (cellulitis) (Infections and infestations) | 1 | 0 | 0 | 0
Infection with unknown ANC: Vagina (Infections and infestations) | 1 | 0 | 0 | 0
Muscle weakness, generalized or specific area (not due to neuropathy): Whole body/generalized (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3 | 0
Partial Thromboplastin Time (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
Pain: Back (General disorders) | 1 | 1 | 0 | 0
Pain: Cardiac/heart (General disorders) | 1 | 0 | 0 | 0
Pain: Chest wall (General disorders) | 1 | 0 | 0 | 0
Pain: External ear (General disorders) | 1 | 0 | 0 | 0
Pain: Face (General disorders) | 1 | 0 | 0 | 0
Pain: Joint (General disorders) | 1 | 0 | 2 | 0
Pain: Middle ear (General disorders) | 1 | 0 | 0 | 0
Pain: Pleura (General disorders) | 1 | 0 | 0 | 0
Pain: Skin (General disorders) | 2 | 1 | 0 | 0
Pain: Tumor pain (General disorders) | 1 | 0 | 1 | 0
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0
Salivary gland changes/saliva (General disorders) | 1 | 3 | 0 | 0
Tumor flare (General disorders) | 1 | 0 | 0 | 0
Urinary frequency/urgency (Renal and urinary disorders) | 1 | 1 | 0 | 0
Vessel injury-vein: Extremity-upper (Vascular disorders) | 1 | 0 | 0 | 0
Vessel injury-vein: IVC (Vascular disorders) | 1 | 0 | 0 | 0
Alkalosis (metabolic or respiratory) (7.35-7.45) (Blood and lymphatic system disorders) | 0 | 1 | 2 | 0
Calcium, ionized-low (hypocalcemia) (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Cholesterol, serum-high (hypercholesteremia) (<200) (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Confusion (General disorders) | 0 | 1 | 1 | 0
Gamma-Glutamyl transpeptidase (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Glomerular filtration rate (Renal and urinary disorders) | 0 | 2 | 2 | 0
Hemorrhage, GI: Lower GI NOS (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Hemorrhage, GU: Stoma (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Hemorrhage, pulmonary/upper respiratory: Bronchus (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Infection (Doc.) with Grade 3/4 ANC: Eye NOS (Infections and infestations) | 0 | 1 | 0 | 0
Infection with normal ANC or Grade 1 or 2 neutrophils: Wound (Infections and infestations) | 0 | 1 | 0 | 0
Left ventricular systolic dysfunction (Cardiac disorders) | 0 | 1 | 0 | 0
Mood alteration: Agitation (General disorders) | 0 | 1 | 1 | 0
Neuropathy: sensory (Nervous system disorders) | 0 | 1 | 0 | 0
Pain - Other (General disorders) | 0 | 2 | 0 | 0
Pain: Bone (General disorders) | 0 | 1 | 0 | 0
Pain: Extremity-limb (General disorders) | 0 | 1 | 0 | 0
Pain: Pain NOS (General disorders) | 0 | 1 | 0 | 0
Pericardial effusion (non-malignant) (Cardiac disorders) | 0 | 2 | 0 | 0
Psychosis (hallucinations/delusions) (Nervous system disorders) | 0 | 1 | 0 | 0
Taste alteration (dysgeusia) (General disorders) | 0 | 1 | 0 | 0
Triglyceride, serum-high (hypertriglyceridemia) (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Ventricular arrhythmia: Ventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Wound complication, non-infectious (General disorders) | 0 | 1 | 0 | 0
Bicarbonate, serum-low (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (General disorders) | 0 | 0 | 1 | 0
Cardiac ischemia/infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Hemorrhoids (General disorders) | 0 | 0 | 1 | 0
Ileus, GI (Gastrointestinal disorders) | 0 | 0 | 1 | 0 — functional obstruction of bowel, i.e., neuroconstipation
Somnolence/depressed level of consciousness (Nervous system disorders) | 0 | 0 | 1 | 0
Proteinuria (neg, trace) (Renal and urinary disorders) | 1 | 1 | 2 | 0
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 0
Fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Lymphatics (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Ocular/Visual - Other (Eye disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-09-06): https://cdn.clinicaltrials.gov/large-docs/89/NCT00573989/Prot_SAP_000.pdf